CLINICAL TRIAL: NCT01005615
Title: Advanced Restoration Therapies in Spinal Cord Injury. AIM1: Patterned FES Ergometry of Arm and Shoulder in Individuals With Spinal Cord Injury
Brief Title: Patterned Functional Electrical Stimulation (FES) Ergometry of Arm and Shoulder in Individuals With Spinal Cord Injury
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding expired and we were unable to gain new funding
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cristina Sadowsky, M.D., Director, Paralysis Restoration Clinic, International Center for Spinal Cord Injury, Kennedy Krieger Institute; Assistant Professor, Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00014481; w81xwh-08-2-0192; W81XWH-09-2-0186
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- No FES Cycling (Sham Comparator)
  Interventions: Device: Non-FES Upper Extremity Exercise
- FES Cycling (Active Comparator)
  Interventions: Device: RT300-SLSA, from Restorative Therapies, Inc.

INTERVENTIONS:
Device: Non-FES Upper Extremity Exercise — While undergoing the non-FES exercise intervention, the subjects will receive a specific, individualized exercise regimen, consisting of strengthening, stretching, splinting and any other therapeutic interventions that do not use electrical stimulation. Than a 1 month washout period,the subjects will remain seated in their primary wheelchair throughout the treatment. The subjects will exercise for 60 minutes/session, three times a week for 4 months.
  Arms: No FES Cycling
Device: RT300-SLSA, from Restorative Therapies, Inc. — They will undergo 4 months of FES assisted upper extremity ergometry followed by 1 month was out period, than by 4 months of a specific, individualized, non FES assisted exercise regimen
  Arms: FES Cycling

SUMMARY:
To determine whether functional electrical stimulation (FES) promotes neurological and physical recovery in patients with spinal cord injury (SCI).

The researchers will investigate the extent of functional recovery in patients with spinal cord injury who receive functional electrical stimulation in the upper extremities compared with patients who do not receive FES.

DETAILED DESCRIPTION:
A randomized, controlled, single-blinded, in-subject controlled (A-B type) trial will be performed in patients with SCI receiving an upper extremities non-FES assisted exercise protocol compared with patients receiving upper extremities ergometry in combination with FES. Neurological and functional outcome measures will be obtained at baseline (time 0), after 1st 4 months of intervention (4 months), after 1 month washout (5 months),after 2nd 4 months intervention (9 months), and 3 month after completing the last intervention (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Male, Female, age 18-55, all ethnic groups
* Spinal Cord Injury, traumatic and non-traumatic
* C1-C6 neurological level
* ASIA class A-B
* Chronic injury > 12 months and < 20 years from the injury
* No upper-extremity electrical stimulation in the previous 4 weeks
* Subjects are medically stable, with no recent (1 month or less) inpatient admission for acute medical or surgical issues
* Baseline physical activity is kept stable
* Pain and antispasticity medications dose are kept stable
* Subjects are legally able to make their own health care decisions

Exclusion Criteria:

* Associated lower motor neuron/peripheral nerve injury in the C1-C6 levels
* Presence of pacemaker
* Presence of cancer
* History of seizures
* Women who are pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina L Sadowsky, MD, Principal Investigator — Kennedy Krieger
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Related Info — http://www.spinalcordrecovery.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was lost to follow up after consent process and 1 Participant was a screen failure neither were assigned which arm/group they would begin in. total number of participants consented were 19 and 17 were assigned.
Period: Intervention 1
Arm/Group | No FES Cycling | FES Cycling
Started | 5 | 12
Completed | 1 | 9
Not Completed | 4 | 3
Period: Washout ()
Arm/Group | No FES Cycling | FES Cycling
Started | 1 | 9
Completed | 1 | 9
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | No FES Cycling | FES Cycling
Started | 1 | 9
Completed | 1 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No FES Cycling | FES Cycling | Total
Number analyzed (Participants) | 5 | 11 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 11 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 11 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Severity of Gleno-humeral Subluxation
Description: This is a routine exam performed to assess shoulder subluxation. The space between the glenoid and head of the humerus can be visualized on plain X-rays and measured, in centimeters, to grade severity. This test is done bilaterally
Time Frame: Baseline
Population: no participants in the no FES cycling arm completed this assessment. 5 participants in the FES cycling arm completed this assessment.
Measure: Mean (Full Range); unit: centimeters
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 0 | 5
centimeters
  Left Side IR |  | 2.2156 [1.569 to 2.789]
  Right Side IR |  | 2.0586 [1.525 to 3.036]

2. Primary Outcome: Severity of Gleno-humeral Subluxation
Description: as for outcome 1
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: centimeters
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 0 | 5
centimeters
  Left Side |  | 2.0146 [1.663 to 2.735]
  Right Side |  | 1.9764 [1.745 to 2.251]

3. Primary Outcome: Severity of Gleno-humeral Subluxation
Description: as for outcome 1
Time Frame: 9 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: centimeters
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 0 | 5
centimeters
  Left Side |  | 2.069 [1.652 to 2.312]
  Right Side |  | 1.997 [1.090 to 3.230]

4. Primary Outcome: Severity of Gleno-humeral Subluxation
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: centimeters
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 0 | 5
centimeters
  Left Side |  | 1.803 [1.421 to 2.161]
  Right Side |  | 1.854 [1.033 to 2.420]

5. Primary Outcome: Modified Ashworth Scale
Description: This is a routine exam performed for people with spinal cord injury.The Modified Ashworth Scale assesses muscle resistance to passive movement. The evaluator moves the joint through the available range of motion and assigns a score from 0-4, where 0 is no tone and 4 is fixed limb (ordinal scale, [44]).Subjects are tested in a seated position preferably in their wheelchairs. The subjects' upper extremity is stabilized by the examiner above and below the joint to be tested. Then the joint is quickly moved through the previously determined subjects' maximum range of motion
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 9
score on a scale
  Baseline | 1 [1 to 1] | 0.333 [0 to 1]
  4th month | 2 [2 to 2] | 0.111 [0 to 1]
  5th month | 3 [3 to 3] | 0.111 [0 to 1]
  9 month | 3 [3 to 3] | 0.333 [0 to 1]
  12 month | 3 [3 to 3] | 0.222 [0 to 2]

6. Primary Outcome: Capabilities of the Upper Extremity (CUE) Test
Description: This is a routine exam performed for people with spinal cord injury.The CUE test is a 32-item interview. It is designed to self-assess upper extremity performance on a 7-point scale (nominal scale, [45]).Subjects are questioned while sitting in their wheelchairs. A brief description of the test will be read to the subjects and then questions asked, one at a time. Subjects will give verbal responses on a 7-point likert scale. total score possible is 0- 225, higher the score better outcome
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Population: Participant did not complete this measure at some time points
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 9
score on a scale
  Baseline: number analyzed (Participants) | 0 | 9
  Baseline |  | 86.55 [32 to 211]
  4th month: number analyzed (Participants) | 0 | 9
  4th month |  | 90.11 [32 to 196]
  5th month: number analyzed (Participants) | 0 | 9
  5th month |  | 97.77 [32 to 210]
  9th month | 76 [76 to 76] | 100.33 [32 to 216]
  12th month | 65 [65 to 65] | 93.22 [32 to 212]

7. Primary Outcome: Jebsen-Taylor Hand Function (JTHF) Test
Description: This is a routine exam performed for people with spinal cord injury.The JTHF test is a 7-item test designed to objectively assess various hand functions and speed of performance (ordinal scale, [46]). Subjects are tested in a seated position, preferably from their wheelchairs, in front of a table. Test items will be laid out on the table and the test conducted per the standardized instructions. The JTHF requires subjects to reach for, lift, and in some cases manipulate small objects. smallest time in seconds mean a better outcome
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Population: Majority of the participants were unable to complete this task
Measure: Mean (Full Range); unit: time in seconds
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 0 | 4
time in seconds
  Baseline: number analyzed (Participants) | 0 | 3
  Baseline |  | 12 [9 to 17]
  4th Month: number analyzed (Participants) | 0 | 3
  4th Month |  | 15 [8 to 28]
  5th Month: number analyzed (Participants) | 0 | 3
  5th Month |  | 15 [8 to 21]
  9th Month |  | 11 [5 to 23]
  12th Month |  | 9 [5 to 17]

8. Primary Outcome: Box and Blocks (BB) Test
Description: This is a routine exam performed for people with spinal cord injury. The BB assesses gross hand function. Subjects are tested in a seated position, preferably from their wheelchairs, in front of a table. Test items will be laid out on the table and the test conducted per the standardized instructions. The BB requires subjects to reach for, lift, and move one inch cubes across a divider inside a wooden box. The amount of time (seconds) subject is able to move around is measured. Higher scores mean better outcome by timed test.
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Population: data was only available for 1 subject in the no FES Cycling and that subject scored a Zero
Measure: Mean (Full Range); unit: seconds
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 4
seconds
  Baseline | 0 [0 to 0] | 36.25 [21 to 53]
  4th Month: number analyzed (Participants) | 1 | 3
  4th Month | 0 [0 to 0] | 42.33 [20 to 58]
  5th Month: number analyzed (Participants) | 1 | 3
  5th Month | 0 [0 to 0] | 39.33 [15 to 60]
  9th Month | 0 [0 to 0] | 38.5 [19 to 59]
  12th month | 0 [0 to 0] | 40 [19 to 56]

9. Secondary Outcome: Action Research Arm (ARA) Test
Description: This is a routine exam performed for people with spinal cord injury.The ARA test observationally assesses upper extremity function .Subjects are tested in a seated position, preferably from their wheelchairs, in front of a table. Test items will be laid out on the table and the test conducted per the standardized instructions. The ARA requires subjects to handle objects differing in size, weight and shape. Score range is from 0-57, higher the number means better outcome overall
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Population: data was only available for 1 subject in the no FES Cycling and that subject scored a Zero
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 4
score on a scale
  Baseline | 0 [0 to 0] | 36.75 [8 to 57]
  4th Month | 0 [0 to 0] | 38 [7 to 57]
  5th Month | 0 [0 to 0] | 38.25 [7 to 57]
  9th Month | 0 [0 to 0] | 34.25 [2 to 57]
  12th Month | 0 [0 to 0] | 36.75 [0 to 57]

10. Secondary Outcome: Range of Motion
Description: This is a routine exam performed for people with spinal cord injury. Subjects are tested in a seated position, preferably in their wheelchairs. The desired joint is isolated and moved through the maximum available range of motion. Once the end range is reached, joint excursion is measured with a goniometer. This measure is to see if you have any active range of motion. 1 is yes to active range of motion and 0 is no range of motion. Having active range of motion is a better outcome
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 9
units on a scale
  Baseline | 1 [1 to 1] | 0.67 [0 to 1]
  4th Month | 1 [1 to 1] | 0.67 [0 to 1]
  5th Month | 1 [1 to 1] | 0.67 [0 to 1]
  9th Month | 1 [1 to 1] | 0.67 [0 to 1]
  12th Month | 1 [1 to 1] | 0.67 [0 to 1]

11. Secondary Outcome: Numerical Rating Scale (NRS).
Description: This is a routine exam performed for people with spinal cord injury. Subjects report how much pain they are having by choosing a number from 0-10, 0 being no pain and 10 being the worst pain
Time Frame: Baseline, 4 months, 5 months, 9 months, 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | No FES Cycling | FES Cycling
Number analyzed (Participants) | 1 | 9
score on a scale
  Baseline | 0 [0 to 0] | 1.67 [0 to 8]
  4th Month | 0 [0 to 0] | 0.78 [0 to 7]
  5th Month | 0 [0 to 0] | 1.89 [0 to 7]
  9th Month | 0 [0 to 0] | 1.56 [0 to 7]
  12th Month | 0 [0 to 0] | 1.11 [0 to 7]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | No FES Cycling | FES Cycling
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT01005615/Prot_SAP_000.pdf